CLINICAL TRIAL: NCT05658731
Title: Cognitive Outcomes After Brain Substructure-informed Radiation Planning in Pediatric Patients
Acronym: CogRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Clark Charitable Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J2255; IRB00331759 (Other: JHM IRB)
Record Dates: First submitted 2022-10-31; First posted 2022-12-21 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Brain Tumor; Head and Neck Cancer
Keywords: radiation therapy; pediatric
MeSH Terms: conditions — Brain Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Stratum A: patients with new diagnosis of brain or head and neck cancer who will be undergoing radiation therapy with substructure informed planning
  Stratum B: patients ≥ 2 years from radiation therapy for brain tumor who underwent standard planning radiation therapy
  Stratum C: healthy controls matched to Stratum A patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stratum A (new diagnosis, substructure informed radiation therapy) (Experimental): Patients will undergo radiation therapy which has been planned according to dose constraints to specific brain substructures.
  Interventions: Radiation: substructure informed planning; Other: Neurocognitive Testing; Diagnostic Test: MRI
- Stratum B (patients ≥ 2 years after standard radiation therapy) (Other): Patients who completed radiation therapy under standard planning procedures ≥ 2 years ago.
  Interventions: Other: Neurocognitive Testing; Diagnostic Test: MRI
- Stratum C (healthy controls matched to Stratum A) (Other): Healthy patients who are matched to Stratum A patients
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Radiation: substructure informed planning — Radiation Therapy with substructure informed planning determined by the PI.
  Arms: Stratum A (new diagnosis, substructure informed radiation therapy)
Other: Neurocognitive Testing — California Verbal Learning Test (CVLT) and other cognition assessments.
  Arms: Stratum A (new diagnosis, substructure informed radiation therapy); Stratum B (patients ≥ 2 years after standard radiation therapy)
Diagnostic Test: MRI — Magnetic resonance imaging (MRI) using whole brain diffusion tensor imaging (DTI) and resting state functional MRI (rsfMRI).

SUMMARY:
The goal of this trial is to determine whether it is possible to minimize radiation dose to parts of the brain that are important for thinking and learning in children who require radiation to treat their tumor, and if this will help reduce neurocognitive (thinking and learning) impairments in these patients.

Patients with newly diagnosed brain or head and neck tumors who are having radiation therapy will have neurocognitive testing and MRI imaging (both research and for regular care) done as part of their participation in the study.

Survivors of childhood brain tumors who completed radiation therapy at least two years before joining the study, and have not had a recurrence, will have neurocognitive testing and research MRIs completed.

Healthy children will also be enrolled and have research MRIs done.

The researchers will use the radiation plan to determine how much radiation was delivered to different parts of the brain. The investigators will use the MRIs to determine how the normal brain is changing after treatment; and how this compares to patients who had standard radiation treatment or who never had a brain tumor. The neurocognitive testing will be compared among different groups to see how different treatment plans affect performance on neurocognitive tests.

ELIGIBILITY:
1. STRATUM A

   1. Eligibility Criteria

      * aged 1 to <26 years of age
      * tumor must be located in the brain or adjacent to the brain including but not limited to nasopharynx, paranasal sinuses and orbit
      * treatment must include radiation therapy (either proton or photon)
      * patients must not have completed radiation therapy
   2. Exclusion Criteria

      * pregnancy
      * patients who are not able to undergo neuro-cognitive testing, including children lacking English comprehension or children with premorbid neurological/neurodevelopmental disorders such as Down's syndrome or autism
2. STRATUM B

   1. Eligibility Criteria

      * diagnosed with a brain tumor at <26 years of age
      * received radiation to the brain as part of therapy
      * time from radiation start to study enrollment is ≥ 2 years
      * there has not been disease recurrence from time of most recent radiation treatment to study enrollment
   2. Exclusion Criteria

      * patients who are not able to undergo neuro-cognitive testing, including children lacking English comprehension or children with premorbid neurological/neurodevelopmental disorders such as Down's syndrome or autism
3. STRATUM C

   1. Eligibility Criteria

      * must be aged 5 to <26 years of age
      * must be able to complete research imaging without sedation
   2. Exclusion Criteria

      * must not have any major psychiatric, neurologic or medical diagnosis

Ages: 1 Year to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 338 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Number of plans that meet substructure-informed planning constraints | 1 month
  Number of plans that meet substructure-informed constraints (per protocol) divided by the total number of plans.

SECONDARY OUTCOMES:
Cumulative incidence of local and distant tumor recurrence | up to 5 years after treatment
  Calculate the cumulative incidence of local and distant tumor recurrence. Local and tumor recurrence is determined by imaging and clinical symptoms.
Fractional anisotropy values | baseline to two years
  This outcome will measure changes in connection strength within brain networks. Fractional anisotropy values range from 0 to 1. Higher numbers are better.
compare the change in California Verbal Learning Test (CVLT) in patients whose radiation plans meet the dose constraints compared to those who do not for all patients in Stratum A. | baseline to 3 years
  Scores are age-standardized and with a mean of 100 and standard deviation of 15. Higher scores are better.
compare the change in NIH toolbox scores in patients whose radiation plans meet the dose constraints compared to those who do not for all patients in Stratum A. | baseline to 5 years
  Scores are age-standardized and with a mean of 100 and standard deviation of 15. Higher scores are better.
characterize longitudinal CVLT scores in survivors of pediatric brain tumor who are ≥ 2 years post radiation | baseline to 5 years
  Scores are age-standardized and with a mean of 100 and standard deviation of 15. Higher scores are better.
characterize longitudinal NIH toolbox scores in survivors of pediatric brain tumor who are ≥ 2 years post radiation | baseline to 5 years
  Scores are age-standardized and with a mean of 100 and standard deviation of 15. Higher scores are better.

CONTACTS AND LOCATIONS:
Overall Officials: Sahaja Acharya, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No